CLINICAL TRIAL: NCT00000902
Title: RAD-1: A Phase I/II Antiretroviral Management Algorithm for Pediatric Subjects of Four-Drug Combination Therapies Based on Prior Antiretroviral Experience
Brief Title: A Study on the Management of Combination Anti-HIV Drug Therapy in HIV-Positive Children With Prior Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 366; 11329 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Zidovudine; Nevirapine; Stavudine; Ritonavir; Lamivudine; RNA, Viral; Anti-HIV Agents; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Nevirapine; Lamivudine; Stavudine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
The purpose of this study is to determine the value of changing anti-HIV medications in children with progressive HIV disease who have received previous treatment.

Plasma viral load (the level of HIV in the blood) is probably most effectively reduced by giving patients anti-HIV drugs which affect the virus at various stages of development. Changing the medications may enhance the results of treatment.

DETAILED DESCRIPTION:
The Master RAD Protocol is based on the concept that optimal suppression of viral load in vivo will be achieved in patients with rapidly progressing or advanced HIV disease (RAD) using antiretroviral combinations inhibiting viral replication at distinct sites of action. Antiretroviral combinations are chosen with the hypothesis that simultaneous change to as many new agents as possible is necessary to maximally reduce plasma viral load.

In this open-label, multicenter study patients are randomized into 1 of 4 groups based on prior antiretroviral experience. Each regimen consists of 4 drugs that include a combination of nucleoside reverse transcriptase inhibitors (stavudine, lamivudine, zidovudine, didanosine, zalcitabine) plus nevirapine (NVP), nelfinavir (NFV), or ritonavir (RTV). Patients must be naive to at least 2 of the 4 drugs in the regimen and at least 1 of the novel drugs must be NVP, NFV, or RTV.

Prior to randomization to a NFV- or RTV-containing regimen, patients are stratified by HIV RNA (greater than or equal to 50,000 or less than 50,000) and must able to receive 2 or more novel drugs.

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he or she:

* Is HIV-positive.
* Is between the ages of 6 months and 21 years (consent of parent or guardian required if under 18).
* Has an HIV blood level above 50,000 copies/mL on 2 consecutive occasions, while taking anti-HIV therapy.
* Has advanced HIV disease or disease progression while receiving 8 weeks or more of continuous unchanged anti-HIV therapy.
* Is able to receive at least one of the following: RTV, NVP, or NFV.

Exclusion Criteria

Your child will not be eligible for this study if he or she:

* Is receiving treatment for a serious bacterial, viral, or opportunistic (HIV-associated) infection within 14 days prior to study entry.
* Has a history of pancreatitis or peripheral neuropathy.
* Has cancer requiring chemotherapy.
* Is allergic to the study medications.
* Is taking certain medications.
* Is pregnant.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 217
Dates: Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kovacs, Study Chair; Sandra Burchett, Study Chair
Locations (62):
- United States (59):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Weinberg A, Kovacs A, Pahwa S, Carey V, Oyomopito R, Mofenson L, Khoury M, Zimmer B, Burchett S. HIV-infected children on HAART reconstitute tetanus-specific T cell responses without booster vaccination. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 688)
- [Background] Frenkel LM, Burchett SK, Aldrovandi GM, Carey V, Oyomopito R, Mahalanibis M, Decker D, Kovacs A. HIV-1 reverse transcriptase (RT) M184V/I improves the rate of suppression of viral replication by salvage therapy. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 463)
- [Background] Kovacs A, Burchett S, Khoury M, Carey V, Pahwa S, McIntosh K, Oyomopito R, Smith E, Mofenson L. Virologic and immunologic responses in children with advanced HIV disease on a new HAART regimen (PACTG 366). 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 684)
- [Background] Weinberg A, Pahwa S, Oyomopito R, Carey VJ, Zimmer B, Mofenson L, Kovacs A, Burchett SK; Pediatric AIDS Clinical Trials Group 366 Team. Antimicrobial-specific cell-mediated immune reconstitution in children with advanced human immunodeficiency virus infection receiving highly active antiretroviral therapy. Clin Infect Dis. 2004 Jul 1;39(1):107-14. doi: 10.1086/420931. Epub 2004 Jun 14. PMID 15206061
- [Result] Saitoh A, Sarles E, Capparelli E, Aweeka F, Kovacs A, Burchett SK, Wiznia A, Nachman S, Fenton T, Spector SA. CYP2B6 genetic variants are associated with nevirapine pharmacokinetics and clinical response in HIV-1-infected children. AIDS. 2007 Oct 18;21(16):2191-9. doi: 10.1097/QAD.0b013e3282ef9695. PMID 18090046
- [Result] EV Capparelli, SK Burchett, A Kovacs, M Khoury, R Oyomopito, L Mofenson, B Zimmer, D Holland. Characterization of the Ritonavir-Nelfinavir Pharmacokinetic Interaction in Pediatric Patients with Advanced HIV Disease Using a Mixed Effects Modeling Approach, Pharmacotherapy, (2003), Abstract 67, Vol.23, No.3, pp.401.
- [Result] S. Burchett, M. Khoury, K. McIntosh, V. Carey, R. Oyomopito, L. Mofenson, E. Smith, A. Kovacs, Viral Load Reduction in Children with Advanced HIV Disease Treated with 4-Drug Antiretroviral Treatment Regimens Including NRTIs, Nevirapine, Nelfinavir and/or Ritonavir, CROI, 2000.